CLINICAL TRIAL: NCT01078077
Title: The Impact of a Topical Vasodilating Cream (When Applied to the Clitoris) on the Female Sexual Experience Using a Standard 7 Part Female Sexual Dysfunction Questionnaire
Brief Title: The Impact of a Topical Vasodilating Cream on Female Sexual Experience
Acronym: TVConFSD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Michael Pelekanos MD (Other)
Collaborators: West Penn Allegheny Health System (Other)
Responsible Party: Sponsor-Investigator, Michael Pelekanos MD, michael pelekanos MD, WPAHS, East Suburban Ob Gyn
Organization: East Suburban Ob Gyn (Other)
Other Study IDs: 10-005
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Female Sexual Dysfunction
Keywords: healthy females ages twentyfive through sixty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if a topical vasodilating cream will improve female sexual experience.

DETAILED DESCRIPTION:
To determine in a placebo controlled double blinded study whether a topically applied vasodilating cream will improve the female sexual response as measured by a standard female sexual dysfunction questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Healthy females ages 25 to sixty sexually active

Exclusion Criteria:

* Neurologic disease, on SSRI's,advanced diabetes, non sexually active, mentally incompetent

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sexually active females from ages 25 to sixty not on SSRI's without neurologic disease able sign and understand informed consent
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: michael j pelekanos, MD, Principal Investigator — east surburban obgyn
Locations (3):
- United States (3):
  - East Suburban Obgyn, Monroeville, Pennsylvania
  - West Penn Allegheny Health Center, Monroeville, Pennsylvania
  - West Penn Hospital Forbes Campus, Monroeville, Pennsylvania